CLINICAL TRIAL: NCT04312087
Title: Lateral Neck Lymph Node Mapping in Papillary Thyroid Carcinoma
Brief Title: Lateral Neck Lymph Node Mapping in Thyroid Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TC-MAP
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; lateral neck lymph node; lymph node mapping; neck dissection; sentinel lymph node
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLND (Experimental): Modified lateral neck dissection (compartment II-V) is performed in all patients.
  Interventions: Procedure: Modified lateral neck lymph node dissection
- SLNB (Experimental): Sentinel lymph node biopsy in the lateral neck is performed. The decision of neck dissection is based on the result of sentinel lymph node biopsy.
  Interventions: Procedure: Lateral neck sentinel lymph node biopsy; Procedure: Modified lateral neck lymph node dissection; Procedure: Super selective lateral neck lymph node dissection

INTERVENTIONS:
Procedure: Lateral neck sentinel lymph node biopsy — Lateral neck sentinel lymph node biopsy is performed in all patients in Arm B.
  Arms: SLNB
Procedure: Modified lateral neck lymph node dissection — Modified lateral neck dissection (compartment II-V) is performed in all patients in Arm A, and some of the patients in Arm B (according to sentinel lymph node biopsy results).
Procedure: Super selective lateral neck lymph node dissection — Super selective lateral neck lymph node dissection is performed in some of the patients in Arm B (according to sentinel lymph node biopsy results).
  Arms: SLNB

SUMMARY:
This study includes papillary thyroid cancer patients who have unpalpable lateral neck lymph nodes but suspicious on ultrasound and/or CT. Carbon nanoparticles is used as the tracer for lateral neck lymph node mapping.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed papillary thyroid cancer
* The maximum diameter of the thyroid cancer <3 cm with enough normal thyroid tissue for tracer injection
* Unpalpable lateral neck lymph nodes
* Ultrasound and CT showed suspected lateral neck lymph nodes <2 cm

Exclusion Criteria:

* Previously treated thyroid cancer
* High risk thyroid cancer (e.g. with severe extra-adenial invasion or extensive lymph node metastasis or poorly differentiated thyroid cancer)
* Patients with distant metastasis

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymph node counts | 1 month after surgery
  Dyed versus undyed lymph node counts in lateral neck compartments

SECONDARY OUTCOMES:
Lymph node metastasis rate | 1 month after surgery
  The rate of lymph node metastasis in lateral neck compartments

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No